CLINICAL TRIAL: NCT05345795
Title: Evaluation of Interstitial Lung Disease Trajectories in Patients With Systemic Sclerosis (SCLEROPIDEVOL Study)
Brief Title: Interstitial Lung Disease Trajectories in Patients With Systemic Sclerosis
Acronym: SCLEROPIDEVOL
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Paul DECKER, MD, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2022PI045
Record Dates: First submitted 2022-04-14; First posted 2022-04-26 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Systemic Sclerosis; Interstitial Lung Disease
MeSH Terms: conditions — Scleroderma, Systemic; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SSc-ILD patients

SUMMARY:
Systemic sclerosis (SSc) is a heterogeneous systemic autoimmune disease with distinct prognosis according to patients. In patients with systemic sclerosis, interstitial lung disease (ILD) concerns almost 50 % of patients and represents the main cause of mortality. Disease course in SSc-ILD is highly variable: patients can experience stable disease, slow or fast progression. Prevention of ILD progression now represents a key objective of SSc-ILD management. The understanding of the course and patterns of SSc-ILD progression is necessary, as reliable prediction tools that allow the stratification of the risk of progression. We aimed to identify the longitudinal trajectories of ILD in SSc patients using latent class mixed models and to examine their associations with SSc characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Patients with systemic sclerosis according to 2013 ACR/EULAR criteria
* Patients with interstitial lung disease on HRCT chest
* Patients with PFT at ILD diagnosis and at least 1 PFT evaluation during follow-up

Exclusion Criteria:

* Patients with an alternative diagnosis of SSc-associated ILD (silicosis, sarcoidosis, lung cancer or other significant lung abnormalities)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with systemic sclerosis-interstitial lung disease
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
FVC change over time | at ILD diagnosis (Day 0) and within 5 years after ILD diagnosis
  evaluation of %predicted FVC values over time using latent class mixed models (LCMM)

SECONDARY OUTCOMES:
DLCO change over time | at ILD diagnosis (Day 0) and within 5 years after ILD diagnosis
  evaluation of %predicted DLCO values over time using latent class mixed models (LCMM)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nancy, Vandœuvre-lès-Nancy, Grand Est, France